CLINICAL TRIAL: NCT00063492
Title: Angiotensinogen Gene and Human Hypertension
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1215; R01HL070048 (NIH)
Record Dates: First submitted 2003-06-30; First posted 2003-07-01 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To determine the role of the angiotensinogen gene in human hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

Essential hypertension affects at least 25 percent of American adults, and it is a primary risk factor for heart failure, stroke, and kidney disease. Many, but not all, studies have shown that variants of the angiotensinogen gene (AGT) affect the risk of hypertension, but association studies conducted to date have been compromised by genetic heterogeneity and by the inherent complexity of hypertension as a phenotype.

DESIGN NARRATIVE:

A comprehensive study of the angiotensinogen (AGT) gene will be conducted in data collected from several large groups of individuals. The investigators will sequence or genotype a 14.4 kb region including AGT in more than 1,600 individuals sampled from populations throughout the world. This will permit them to explore fully the extent of allelic heterogeneity, haplotype variation, and potential for population stratification in the AGT gene. Approximately 600 of these individuals are clinically uncharacterized and will represent a broad range of worldwide human variation. Another 500 subjects are members of 40 Utah pedigrees that are part of the Centre d'Etude du Polymorphisme Humain (CEPH) collection. These unique families have been heavily characterized genetically, and they are now being phenotyped for variables that include anthropometrics, blood chemistries, blood pressure measures, and plasma and urinary angiotensinogen. They will address the issue of genetic heterogeneity by testing associations between multi-SNP AGT haplotypes, angiotensinogen levels, and blood pressure. In addition, linkage disequilibrium patterns will be assessed to determine the density and nature of SNPs best suited for localizing a gene underlying a complex trait. They will address the issue of phenotypic heterogeneity in hypertension by performing extensive SNP typing on a set of 400 hypertensives and 100 normotensives collected by Dr. Gordon Williams. These clinically well-characterized subjects have been tested for their response to infused angiotensin-II under high and low sodium intake. This direct probe provides a hypertension endophenotype that is closer to the function of the AGT gene, yielding a more realistic and informative assessment of the relationship between AGT haplotype variation and hypertension risk. A phylogenetic analysis of AGT sequence variation in the worldwide sample will help to assess population stratification in association studies. In addition, this sample will allow testing the hypothesis that the ancestral T235 AGT allele provided a selective advantage in the sodium-poor environment of sub-Saharan Africa. The results of this analysis may help to explain why African-Americans have elevated rates of hypertension. In summary, the extensive analysis of AGT variation in more than 1,600 subjects will clarify the role of this gene in essential hypertension and will test specific hypotheses about the evolution of AGT.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Jorde — University of Utah

REFERENCES:
- [Background] Nakajima T, Wooding S, Satta Y, Jinnai N, Goto S, Hayasaka I, Saitou N, Guan-Jun J, Tokunaga K, Jorde LB, Emi M, Inoue I. Evidence for natural selection in the HAVCR1 gene: high degree of amino-acid variability in the mucin domain of human HAVCR1 protein. Genes Immun. 2005 Aug;6(5):398-406. doi: 10.1038/sj.gene.6364215. PMID 15889130